CLINICAL TRIAL: NCT02145546
Title: Antiarrhythmic Drugs Assessment in Preventing Atrial Fibrillation
Acronym: ADA-PAF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Medtronic (Shanghai) Management Co. Ltd. (Industry); Beijing CTSmed Co. Ltd (Unknown)
Responsible Party: Principal Investigator, Yi-Gang Li, Chief Physician, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2013-013-2
Record Dates: First submitted 2014-04-02; First posted 2014-05-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Atrial Fibrillation
Keywords: Pacing dependent; Atrial Fibrillation; Amiodarone; Propafenone; Sotalol; AF burden
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone; Propafenone; Sotalol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Amiodarone (Experimental): Patient will take Amiodarone orally
  Interventions: Drug: Amiodarone
- Sotalol (Experimental): Patients will take sotalol orally
  Interventions: Drug: Sotalol
- Propafenone (Experimental): Patients will take propafenone orally
  Interventions: Drug: Propafenone
- Control (No Intervention): Patients will take no antiarrhythmic drugs except β-blocker

INTERVENTIONS:
Drug: Amiodarone — Amiodarone: 200mg three times a day for two weeks, then change to 200mg per day for the rest of the study.
  Other Names: cordarone; pacerone; aratac; arycor; atlansil; tachyra
  Arms: Amiodarone
Drug: Propafenone — 150mg per 8 hours, 3 times per day
  Other Names: rythmol SR; rytmonorm
  Arms: Propafenone
Drug: Sotalol — 80mg twice per day.
  Other Names: betapace; betapace AF; sotalex; sotacor
  Arms: Sotalol

SUMMARY:
The current evidences indicate that ~30% patients with sick sinus syndrome(SSS) would develop persistent atrial fibrillation (AF) after a long term pacing therapy. However, the accurate influence of antiarrhythmic drugs on the AF is still not well defined. The purpose of the study is to assess the therapeutic effects of various antiarrhythmic drugs (Amiodarone, Sotalol and Propafenone) on the long term management of AF in SSS patients with AF, including the reduced AF burden (duration and episodes) and persistent AF free survival rate. All patients will be followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* sick sinus syndrome with pacemaker Class I or Class IIa indication
* has a pacemaker which can provide the daily AF burden monitor record for at least 28 days
* has at AF record in the past 6 months, the valid AF record includes any of

  1. at least one 30 seconds AF holter record
  2. at least one 15 seconds 12-ECG record
  3. at least 5 minutes long AF episodes record from pacemakers
* able and willing to give informed consent

Exclusion Criteria:

* will have cardiac surgery in the next 6 month or in the waiting list of heart transplantation
* NYHA Class III or IV
* LVEF <50%
* Reversible AF, such as AF caused by hyperthyroidism or severe postoperative atrial fibrillation
* Persistence AF
* Expected life expectancy less than 1 year
* Planned to be pregnant or be in the feeding period in the next year
* Non-stable, decompensated heart failure
* Allergy to Amiodarone, Propafenone or Sotalol
* Cancer
* Clear liver damage ( ALT and/or AST > 2*normal limit)
* Patients with cardiogenic shock history
* Be in the treatment of Amiodarone for more than 3 months or less than 3 months with Amiodarone wash out period less than 30 days
* Coronary artery disease (CHD), cardiomyopathy, severe valvular heart disease, severe obstructive pulmonary disease (COPD), long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Average AF burden in minutes per day | monthly up to 12 months
  Long term usages of test drug reduce AF burden, including the number and accumulated total time of AF per day.
Persistent AF free survival rate | monthly up to12 months
  Long term usages of test drugs reduce the occurence of the persistent AF ( the persistent AF survival rate)。

SECONDARY OUTCOMES:
Left ventricular function | 0months, 6months and 12 months
  LVEF(Simpson), LV volume, diastolic function (E/A ), tricuspid regurgitation, Left atrial size and volume
SF-36 health survey | 0 months, 6 months and 12 months
  SF-36 health survey
comorbidity and mortality | 6 months and 12 months
  The rate of stroke, infarction, heart failure, rehospitalization and cardiovascular and total mortality rate.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Gang Li, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiaotong University School of Medicne
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicne, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] OSTRANDER LD Jr, BRANDT RL, KJELSBERG MO, EPSTEIN FH. ELECTROCARDIOGRAPHIC FINDINGS AMONG THE ADULT POPULATION OF A TOTAL NATURAL COMMUNITY, TECUMSEH, MICHIGAN. Circulation. 1965 Jun;31:888-98. doi: 10.1161/01.cir.31.6.888. No abstract available. PMID 14297523
- [Background] Zhou ZQ, Hu DY, Chen J, Zhang RH, Li KB, Zhao XL. [An epidemiological survey of atrial fibrillation in China]. Zhonghua Nei Ke Za Zhi. 2004 Jul;43(7):491-4. Chinese. PMID 15312400
- [Background] Siu CW, Jim MH, Zhang X, Chan YH, Pong V, Kwok J, Kung AW, Lau CP, Tse HF. Comparison of atrial fibrillation recurrence rates after successful electrical cardioversion in patients with hyperthyroidism-induced versus non-hyperthyroidism-induced persistent atrial fibrillation. Am J Cardiol. 2009 Feb 15;103(4):540-3. doi: 10.1016/j.amjcard.2008.10.019. Epub 2008 Dec 25. PMID 19195517
- [Background] Singh BN, Singh SN, Reda DJ, Tang XC, Lopez B, Harris CL, Fletcher RD, Sharma SC, Atwood JE, Jacobson AK, Lewis HD Jr, Raisch DW, Ezekowitz MD; Sotalol Amiodarone Atrial Fibrillation Efficacy Trial (SAFE-T) Investigators. Amiodarone versus sotalol for atrial fibrillation. N Engl J Med. 2005 May 5;352(18):1861-72. doi: 10.1056/NEJMoa041705. PMID 15872201
- [Background] Roy D, Talajic M, Dorian P, Connolly S, Eisenberg MJ, Green M, Kus T, Lambert J, Dubuc M, Gagne P, Nattel S, Thibault B. Amiodarone to prevent recurrence of atrial fibrillation. Canadian Trial of Atrial Fibrillation Investigators. N Engl J Med. 2000 Mar 30;342(13):913-20. doi: 10.1056/NEJM200003303421302. PMID 10738049
- [Background] Pritchett EL, Page RL, Carlson M, Undesser K, Fava G; Rythmol Atrial Fibrillation Trial (RAFT) Investigators. Efficacy and safety of sustained-release propafenone (propafenone SR) for patients with atrial fibrillation. Am J Cardiol. 2003 Oct 15;92(8):941-6. doi: 10.1016/s0002-9149(03)00974-3. PMID 14556870
- [Background] Israel CW. Analysis of mode switching algorithms in dual chamber pacemakers. Pacing Clin Electrophysiol. 2002 Mar;25(3):380-93. doi: 10.1046/j.1460-9592.2002.00380.x. PMID 11990674
- [Background] Passman RS, Weinberg KM, Freher M, Denes P, Schaechter A, Goldberger JJ, Kadish AH. Accuracy of mode switch algorithms for detection of atrial tachyarrhythmias. J Cardiovasc Electrophysiol. 2004 Jul;15(7):773-7. doi: 10.1046/j.1540-8167.2004.03537.x. PMID 15250860
- [Background] Kaufman ES, Israel CW, Nair GM, Armaganijan L, Divakaramenon S, Mairesse GH, Brandes A, Crystal E, Costantini O, Sandhu RK, Parkash R, Connolly SJ, Hohnloser SH, Healey JS; ASSERT Steering Committee and Investigators. Positive predictive value of device-detected atrial high-rate episodes at different rates and durations: an analysis from ASSERT. Heart Rhythm. 2012 Aug;9(8):1241-6. doi: 10.1016/j.hrthm.2012.03.017. Epub 2012 Mar 20. PMID 22440154
- [Background] Nowak B, McMeekin J, Knops M, Wille B, Schroder E, Moro C, Oelher M, Castellanos E, Coutu B, Petersen B, Pfeil W, Kreuzer J; Stored EGM in PulsarMax II and Discovery II Study Group. Validation of dual-chamber pacemaker diagnostic data using dual-channel stored electrograms. Pacing Clin Electrophysiol. 2005 Jul;28(7):620-9. doi: 10.1111/j.1540-8159.2005.00159.x. PMID 16008796
- [Background] Charles D. Swerdlow, Jeffrey M. Gillberg, Paul Khairy, Textbook, Clinical Cardiac Pacing, Defibrillation and Resynchronization Therapy, Chapter 3, Sensing and Detection, page 146.